CLINICAL TRIAL: NCT06776796
Title: A Pilot Randomized Controlled Trial to Test the Efficacy of a Brief Alcohol Intervention Among College Students
Brief Title: Testing the Efficacy of a Brief Alcohol Intervention Among College Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Georgia State University (Other)
Responsible Party: Principal Investigator, Amanda Gilmore, Associate Professor and PhD Director, Department of Health Policy & Behavioral Sciences Director, National Center for Sexual Violence Prevention, Georgia State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: H24001
Record Dates: First submitted 2025-01-08; First posted 2025-01-15 (Actual); Last update posted 2025-01-15 (Actual); Status verified 2025-01

CONDITIONS: Alcohol Use; Personalized Normative Feedback
MeSH Terms: conditions — Alcohol Drinking | interventions — Ethanol; Mental Health

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participants will be masked to intervention conditions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Online Personalized Normative Feedback Intervention Targeting Alcohol Misuse (Experimental): This is an integrated social norms-based personalized feedback intervention for college students targeting alcohol misuse. It is tailored by the identities chosen by participants including gender, race/ethnicity, and sexual orientation. The intervention is a modified version of an existing evidence-based program, the Brief Alcohol Screening and Intervention for College Students (BASICS) (Dimeff, et. al, 1999).
  Interventions: Behavioral: Online Personalized Normative Feedback Intervention Targeting Alcohol Misuse
- Mental Health and Substance Use Resources (Placebo Comparator): Participants were directed to a website where information regarding mental health and substance use may be found.
  Interventions: Behavioral: Mental Health and Substance Use Resources

INTERVENTIONS:
Behavioral: Online Personalized Normative Feedback Intervention Targeting Alcohol Misuse — This is an integrated social norms-based personalized feedback intervention for college students targeting alcohol misuse. It is tailored by the identities chosen by participants including gender, race/ethnicity, and sexual orientation. The intervention is a modified version of an existing evidence-based program, the Brief Alcohol Screening and Intervention for College Students (BASICS) (Dimeff, et. al, 1999).
  Arms: Online Personalized Normative Feedback Intervention Targeting Alcohol Misuse
Behavioral: Mental Health and Substance Use Resources — Participants were directed to a website where information regarding mental health and substance use may be found.
  Arms: Mental Health and Substance Use Resources

SUMMARY:
Individuals will be recruited to participate in a randomized controlled trial to test the efficacy of a prevention program aimed at reducing alcohol use among college students. If randomized to the intervention, participants will view personalized content based on their alcohol use and chosen identity and learn about various topics related to alcohol use, including ways to reduce their use. Control participants will be directed to a website where information regarding mental health and substance use may be found. Baseline mental health, alcohol use, and related constructs will be assessed. Participants will complete a 3-month follow-up survey to assess the efficacy of the tool in symptom reduction.

DETAILED DESCRIPTION:
Students will be recruited by campus flyers, social media, and a registrar list to participate in a randomized controlled trial (RCT) to test the efficacy of a prevention program aimed at reducing alcohol use among college students. Participants will also be recruited from a list of students who completed the Panthers4Life community needs assessment. Interested students will first complete a screener to determine eligibility (i.e., enrolled GSU student, 18-25 years of age, identifies as Black, White and LGBTQA+, Latine/a/o or Hispanic, and engaged in heavy episodic drinking at least once in the past month). Individuals who identify their sex at birth to be intersex or who identify themselves to be both heterosexual and gender diverse (Transgender, Genderqueer, Gender non-conforming, Non-binary, Androgynous, and Two-spirit) will be excluded due to the lack of normative data about these groups. Eligible participants will immediately be given the informed consent and asked to complete a baseline survey (15 minutes). In the baseline survey, participants will select identity group(s) they most identify with and select identity group(s) they would like to receive personalized normative feedback about. Participants will then be randomized to either complete a brief online intervention (treatment group) or view website information about substance use and mental health (control group).

If randomized to the intervention, participants will complete an intervention in Qualtrics Survey Platform that takes approximately 15 minutes to complete. They will view personalized content based on their alcohol use and chosen identity (e.g., if a participant chooses woman and LGBQA+ they will receive personalized normative feedback for women LGBQA+ students at GSU) and learn about various topics related to alcohol use, including ways to reduce their use. The intervention is a modified version of an existing evidence-based program, the Brief Alcohol Screening and Intervention for College Students (BASICS).

Participants assigned the control condition will be directed to a website where information regarding mental health and substance use may be found.

In both groups, the investigators will assess baseline mental health, alcohol use, and related constructs. Both groups will also be asked to complete a 3-month follow-up survey to assess the efficacy of the tool in symptom reduction. Cultural acceptability will also be assessed to determine if cultural adaptations are needed to enhance efficacy among groups represented in our sample. Participants will be compensated up to $30 in Amazon gift cards for their time ($15 for the baseline survey and $15 for the 3-month follow up).

ELIGIBILITY:
Inclusion Criteria:

* 18-25 years old
* Current student at university of study
* Valid email address at university of study
* Identifies as Black, White and LGBTQA+, Latine/a/o or Hispanic,
* Endorse engaging in heavy episodic drinking at least once in the past month on the screening survey

Exclusion Criteria:

• Individuals who identify their sex at birth as intersex or who identify as both heterosexual and gender diverse (Transgender, Genderqueer, Gender non-conforming, Non-binary, Androgynous, and Two-spirit) will be excluded due to the lack of normative data about these groups.

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 461 (Actual)
Dates: Start 2023-08-23 (Actual); Primary Completion 2024-01-21 (Actual); Study Completion 2024-01-21 (Actual)

PRIMARY OUTCOMES:
Changes in Alcohol use | Baseline and 3-months
  Number of drinks will be assessed using the daily drinking questionnaire. Higher scores indicate higher alcohol use.

CONTACTS AND LOCATIONS:
Locations (1):
- Georiga State University, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Gilmore AK, Leone RM, Reuben K, Garner JB, Flowers N, Chipman T, Patton EE, Capobianco J, Zong ZY, Stappenbeck CA, Ellis JR, Fortson K, Mullican KN, Larimer M. Pilot randomized controlled trial of a tailored personalized normative feedback intervention for college student alcohol use. Drug Alcohol Depend. 2025 Oct 1;275:112824. doi: 10.1016/j.drugalcdep.2025.112824. Epub 2025 Aug 8. PMID 40834655

DOCUMENTS (1):
  • Informed Consent Form (2023-06-21): https://cdn.clinicaltrials.gov/large-docs/96/NCT06776796/ICF_000.pdf